CLINICAL TRIAL: NCT03110874
Title: A Multi-center, Randomized, Interventional, Open, Phase Ⅳ Clinical Trial on Education Method of Fluterol® Inhalation Capsule 250/50 μg Inhaler for Asthma Control in Patients With Partly Controlled Asthma
Brief Title: Clinical Trial on Education Method of Fluterol® Inhalation Inhaler for Asthma Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM-FLU-401
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (one-way education) (Experimental): Experimental group (one-way education)
  * Fluterol Inhalation Capsule (fluticasone propionate 250 μg, salmeterol xinafoate 72.5 μg)
  * video based education
  Interventions: Drug: one-way education
- Control group(two-way education) (Active Comparator): Control group(two-way education)
  * Fluterol Inhalation Capsule (fluticasone propionate 250 μg, salmeterol xinafoate 72.5 μg)
  * direct education
  Interventions: Drug: two-way education

INTERVENTIONS:
Drug: one-way education — 'Fluterol Inhalation Capsule(fluticasone propionate 250 μg, salmeterol xinafoate 72.5 μg) : one-way education'
  Other Names: video based education
  Arms: Experimental group (one-way education)
Drug: two-way education — 'Fluterol Inhalation Capsule(fluticasone propionate 250 μg, salmeterol xinafoate 72.5 μg) : two-way education'
  Other Names: direct education
  Arms: Control group(two-way education)

SUMMARY:
A multi-center, randomized, open, non-inferiority, Phase 4 study

DETAILED DESCRIPTION:
A Multi-center, Randomized, Interventional, Open, Phase Ⅳ Clinical Trial on Education Method of Fluterol® Inhalation Capsule 250/50 μg Inhaler for Asthma Control in Patients with Partly Controlled Asthma

ELIGIBILITY:
Inclusion Criteria:

1. Adult at the age of 19 or older.
2. Patient with partially controlled asthma (Asthma Control Test score 16~24)
3. Written informed consent to study participation.

Exclusion Criteria:

1. History of hypersensitivity reactions to the investigational product (Fluterol®) or any of its component.
2. Cardiac tachyarrhythmia.
3. contreated respiratory fungal, bacterial, or tuberculous infection.
4. Moderate to severe bronchiectasis
5. Planned use of the investigational product (Fluterol®) as primary treatment for patients with status asthmaticus, patients with an asthmatic crisis*, or patients with chronic obstructive pulmonary disease requiring intensive treatment.

   * Asthmatic crisis: acute exacerbation of asthma meeting at least one of the followings.
   * Asthma related emergency room visit or hospitalization within 2 weeks prior to screening.
   * Administration of systemic steroids within 2 weeks prior to screening.
   * Inhalation of rescue medication at least 10 times/day for the treatment of acute exacerbation of asthmatic symptoms within 2 weeks prior to screening.
6. Administration of systemic steroids within 2 weeks prior to screening.
7. Hypersensitivity reactions to lactose and milk.
8. Pregnant and lactating women or women who are planning to be pregnant or who are unwilling to use appropriate methods of contraception during the study.
9. Previous use of the investigational product (Fluterol®) or a similar inhaler (Onbrez, Spiriva) at least once.
10. Participation in another clinical study for drugs or medical devices to receive the investigational product or undergo a procedure using the investigational device within 4 weeks prior to participation in this study.
11. Individual considered by the he investigator to be inappropriate for study participation due to other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Percent change in Forced expiratory volume 1 sec (% prediction) at Week 12 from baseline in each group. | Week 12
  method of assessment:Forced expiratory volume

SECONDARY OUTCOMES:
percent change in Forced expiratory volume 1 sec (% prediction) at Week 4 from baseline in each group. | Week 4
  method of assessment:Forced expiratory volume
Change in asthma control (ACT) at Weeks 4 and 12 from baseline in each group. | Weeks 4 and 12
  method of assessment: Check list
Change in inhaler technique score at Weeks 4 and 12 from baseline in each group | Weeks 4 and 12
  method of assessment: Check list
Number of critical errors at Weeks 4 and 12 in each group. | Weeks 4 and 12
  method of assessment: Check list
Proportion of subjects with optimal inhaler technique at Weeks 4 and 12 in each group. | Weeks 4 and 12
  method of assessment: Check list
Satisfaction for the inhalation drug at Weeks 4 and 12 in each group (FSI-10 score). | Weeks 4 and 12
  method of assessment: Check list
Adherence rate (%) at Weeks 4 and 12 in each group. | Weeks 4 and 12
  method of assessment: drug administration calculation
Safety endpoint:AEs(adverse events), vital signs, incidence rate of acute exacerbation. | baseline(day1),weeks 4 and weeks12
  occur frequency of adverse events and incidence rate of acute in each group, vital signs: blood pressure and pulse

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Whui Choi, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine

IPD SHARING:
Plan to Share IPD: Undecided